CLINICAL TRIAL: NCT02658357
Title: Study in Stabilized Schizophrenic Patients to Evaluate the Pharmacokinetics of Risperidone and 9-Hydroxy (OH)-Risperidone When Risperidone is Administered From a Polyurethane Implant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braeburn Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB-PK-103
Record Dates: First submitted 2016-01-07; First posted 2016-01-18 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia; Schizo-affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 600 mg (Experimental): Two, 300 mg Risperidone Implants
  Interventions: Drug: Risperidone Implant
- 900 mg (Experimental): Three, 300 mg Risperidone Implants
  Interventions: Drug: Risperidone Implant

INTERVENTIONS:
Drug: Risperidone Implant

SUMMARY:
The study will be a 6-month, open-label, multiple center study in approximately 50 stable subjects diagnosed with schizophrenia or schizoaffective disorder to evaluate the safety, tolerability, and pharmacokinetics of Risperidone and 9-OH-Risperidone following implantation of two or three, 300 mg Risperidone Implants.

DETAILED DESCRIPTION:
The study will be a 6-month, open-label, study in approximately 50 stable subjects diagnosed with schizophrenia or schizoaffective disorder to evaluate the safety, tolerability, and pharmacokinetics of Risperidone and 9-OH-Risperidone following implantation of two or three, 300 mg Risperidone Implants.

Subjects who are diagnosed with schizophrenia or schizoaffective disorder according to DSM-V and are stable on a daily 4 mg oral dose of Risperidone for at least 8 weeks will be recruited into the study.

Subjects stable on a 4 mg oral dose of Risperidone will be implanted with two or three, 300 mg, Risperidone Implants. All implants will be placed in the inner aspect of the upper arm. Plasma concentrations of Risperidone and the active moiety will be measured prior to placement of the Risperidone Implants, throughout the implantation period, and after re-converting to oral Risperidone following the removal of the Risperidone Implants.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (and/or a subject's authorized legal representative) has provided written informed consent
2. Patient meets the following criteria:

   * Outpatient status
   * PANSS Total Score ≤ 80 at screening and if PANSS score at baseline is ≥ 20% change from screening, the patients cannot participate in the study.
   * A score of ≤ 3 on the following PANSS items:

     * Conceptual disorganization
     * Suspiciousness
     * Hallucinatory behavior
     * Unusual thought content
3. Subject is male or female between 18 to 60 years of age
4. Subject has a diagnosis of schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria

Exclusion Criteria:

1. Hospitalized or required acute crisis intervention for symptom exacerbation in the 60 days prior to admission as determined by the Investigator
2. Subject has a history of suicide attempt in the last year, or in the opinion of the investigator is currently at imminent risk of suicide
3. Has a current or recent (within 12 months) DSM-V diagnosis of moderate or severe substance use disorder (except for tobacco use disorder) or has a positive urine drug screen for prohibited substances at screening.
4. Have impaired hepatic (ALT/AST >1.5 times higher than the upper limit of normal) or renal function (eGFR<50 mL/min)
5. Previously defined hypersensitivity to Risperidone
6. History of neuromalignant syndrome (NMS)
7. Electroconvulsive therapy within 6 months of admission
8. Requires current use of agents that are strong inhibitors and inducers of cytochrome P450 2D6

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Segal Institute for Clinical Research 1201 North 37th Avenue, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The product was sold to another company prior to data analysis. The new company closed before the results were completed, so no results are available for this study
Groups:
- 600 mg: Two, 300 mg Risperidone Implants
  Risperidone Implant
- 900 mg: Three, 300 mg Risperidone Implants
  Risperidone Implant
Period: Overall Study
Arm/Group | 600 mg | 900 mg
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The product was sold to another company prior to data analysis. The new company closed before the results were completed, so no results are available for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 600 mg | 900 mg | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for Active Moiety, 9-hydroxy-risperidone and Risperidone
Time Frame: 6 months
Population: as for baseline characteristics
Arm/Group | 600 mg | 900 mg
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Cmax for Active Moiety, 9-hydroxy-risperidone and Risperidone
Time Frame: 6 months
Population: as for baseline characteristics
Arm/Group | 600 mg | 900 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Safety and Efficacy of a Risperidone Implant as Assessed by the Positive and Negative Syndrome Scale (PANSS)
Time Frame: 12 months
Population: as for baseline characteristics
Arm/Group | 600 mg | 900 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: The product was sold to another company prior to data analysis. The new company closed before the results were completed, so no results are available for this study.
Arm/Group | 600 mg | 900 mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The product was sold to another company prior to data analysis. The new company closed before the results were completed, so no results are available for this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT02658357/Prot_SAP_000.pdf